CLINICAL TRIAL: NCT03336177
Title: Understanding Low Gynecological Cancer Delay and Help-seeking Behavior in Older Patients. Qualitative Approach
Brief Title: Understanding Low Gynecological Cancer Delay and Help-seeking Behavior in Older Patients.
Acronym: CODEGY65
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01574-49
Record Dates: First submitted 2017-10-19; First posted 2017-11-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Gynecologic Cancer; Symptoms and Signs; Aged
Keywords: gynecology; cancer; aged; delay; help-seeking behavior; qualitative research; semiopragmatic analysis; psychodynamic analysis
MeSH Terms: conditions — Signs and Symptoms; Neoplasms; Help-Seeking Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-structured face to face interviews. — Patients will be interviewed by open-ended questions face to face concerning their past experiences. The recorded interview will be transcribed and analyzed by psychodynamic and semio-pragmatic approach.

SUMMARY:
Systematic screening for cervical cancer stops in France at 65 years old. The incidence of certain types of gynecological neoplasia increases with age (endometrium, vulva). Diagnosis delay of 8 months has been described for uterine cancer and longer delays for vulvar cancer.

The aim of our study is to understand help-seeking behavior and its delay for this type of cancer among patients older than 65.

DETAILED DESCRIPTION:
Our study assess the reasons for which the patient took time to go to the doctor despite of their symptoms. We use a qualitative methodology. Our study categorizes lived experiences, recorded in semistructured interview transcripts. We use psychodynamic and semiopragmatic analyses of the discourse to obtain hypotheses about possible reasons of the delay in the help-seeking process."

ELIGIBILITY:
Inclusion Criteria:

* Women of 65 years or more treated or followed at Lorraine Institute of Oncology
* Diagnosed after 65 years or later of a low gynecological cancer
* Without diagnosis of dementia
* Retained ability to express by herself without assistance
* Affiliated to public health system
* Informed and having expressed her non-opposition

Exclusion Criteria:

* Women under 65 or diagnosed before being 65 of a low gynecological cancer
* Diagnosed of dementia
* No longer to express herself
* Patient deprived of freedom

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Women of 65 years or more treated or followed at Lorraine Institute of Oncology Diagnosed after 65 years or later of a low gynecological cancer
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Experience of help-seeking period for low gynecological cancers. | 1 day
  Qualitative interview performed at one occasion where the patient describes the experience of the help seeking period she has passed through.

SECONDARY OUTCOMES:
Motivators and barriers to help-seeking for low gynecological cancers. | 1 day
  qualitative methodology using verbal data analysis of semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: MARCHAL FREDERIC, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine (ICL), Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No